CLINICAL TRIAL: NCT05161819
Title: Use Repetitive Transcranial Magnetic Stimulation to Treat Somatic Symptom Disorder: A Randomized Double-blind Sham-controlled Crossover Study
Brief Title: Use Repetitive Transcranial Magnetic Stimulation to Treat Somatic Symptom Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 202109065DINC
Record Dates: First submitted 2021-12-05; First posted 2021-12-17 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Somatic Symptom Disorder
Keywords: somatic symptom disorder; repetitive transcranial magnetic stimulation; dorsolateral prefrontal cortex; somatic distress; health anxiety
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-frequency rTMS at left DLPFC (Experimental): Receive an rTMS course with high-frequency stimulation at left DLPFC
  Interventions: Device: Repetitive transcranial magnetic stimulation
- High-frequency sham stimulation at left DLPFC (Sham Comparator): Receive an sham rTMS course with high-frequency stimulation at left DLPFC with the sham coil
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation — High-frequency stimulation (10Hz), 120% motor threshold, 40 trains, 1600 pulses
  Arms: High-frequency rTMS at left DLPFC
Device: Sham stimulation — High-frequency stimulation (10Hz), 120% motor threshold, 40 trains, 1600 pulses (with sham coil)
  Arms: High-frequency sham stimulation at left DLPFC

SUMMARY:
This is a randomized double-blind sham-controlled crossover study; the interventions are high-frequency rTMS stimulation on left DLPFC and sham control. The study population is the patient with somatic symptom disorder. The primary outcomes are somatic distress and health anxiety.

DETAILED DESCRIPTION:
Somatic symptom disorder (SSD) is a psychiatric diagnosis featured with somatic distress and health anxiety. It is overlapped with functional disorders. Whether it has effective treatment is a clinically important issue. Current evidence indicates that pharmacotherapy and psychotherapy are both helpful for SSD. Among other treatment options, repetitive transcranial magnetic stimulation (rTMS) is attached important in psychiatric field; it can cause activation or inhibition of specific brain regions via magnetic stimulation. Previous studies have disclosed that rTMS is helpful for depression, obsessive-compulsive disorder, post-stroke rehabilitation, etc. Regarding functional disorders, fibromyalgia has been found to be benefited from rTMS; the effective approaches include giving high-frequency stimulation on left M1 and dorsolateral prefrontal cortex (DLPFC). Chronic tinnitus was also found to have response to rTMS. SSD and fibromyalgia are highly overlapped; SSD and depression are often comorbid. Therefore, SSD may also be benefited from left DLPFC high-frequency stimulation. Our previous study revealed that dysfunction of anterior cingulate cortex (ACC) is associated with persistent interference of the somatic discomforts; stimulation on DLPFC can cause ACC activation. This study program was designed based on the above information. It is a randomized double-blind sham-controlled crossover study; the interventions are high-frequency rTMS stimulation on left DLPFC and sham control. The primary outcomes are somatic distress and health anxiety. There is not study about rTMS on SSD in literature; the investigators expect this study to be able to provide more understanding on this field.

ELIGIBILITY:
Inclusion Criteria:

* Patient with somatic symptom disorder (confirmed by psychiatrists)
* Age 20-70

Exclusion Criteria:

* Having psychotic symptoms or cognitive impairment
* Having potentially lethal illness
* Using cardiac pacemakers or defibrillators
* Currently pregnant or having plans to become pregnant within the next three months
* Received rTMS treatment within three months
* Cannot read the questionnaires by oneself
* Having to take the following medications persistently: bupropion >300 mg/day、TCA、clozapine、chlorpromazine、foscarnet、ganciclovir、ritonavir、theophylline

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Scores of Patient Health Questionnaire-15 (PHQ-15) | Week 3 (comparing with the data in week 0) of the two sections (rTMS and sham)
  Measurement of somatic distress. Score range is 0 to 30; higher score means more severe somatic distress
Scores of Health Anxiety Questionnaire (HAQ) | Week 3 (comparing with the data in week 0) of the two sections (rTMS and sham)
  Measurement of health anxiety. Score range is 0 to 63; higher score means more severe health anxiety

SECONDARY OUTCOMES:
Scores of Patient Health Questionnaire-15 (PHQ-15) | Week 1, 2 (comparing with the data in week 0) of the two sections (rTMS and sham)
  Measurement of somatic distress. Score range is 0 to 30; higher score means more severe somatic distress
Scores of Health Anxiety Questionnaire (HAQ) | Week 1, 2 (comparing with the data in week 0) of the two sections (rTMS and sham)
  Measurement of health anxiety. Score range is 0 to 63; higher score means more severe health anxiety
Scores of Beck Depression Inventory-II (BDI-II) | Week 1, 2, 3 (comparing with the data in week 0) of the two sections (rTMS and sham)
  Measurement of depression. Score range is 0 to 63; higher score means more severe depression
Scores of Beck Anxiety Inventory (BAI) | Week 1, 2, 3 (comparing with the data in week 0) of the two sections (rTMS and sham)
  Measurement of anxiety. Score range is 0 to 63; higher score means more severe anxiety
Scores of Cognitions About Body and Health Questionnaire (CABAH) | Week 1, 2, 3 (comparing with the data in week 0) of the two sections (rTMS and sham)
  Measurement of cognitions about health. Score range is 0 to 117; higher score means more severe cognitive distortion about health
Heart rate variability | Week 1, 2, 3 (comparing with the data in week 0) of the two sections (rTMS and sham)
  Measurement of parasympathetic activity
Skin conductance | Week 1, 2, 3 (comparing with the data in week 0) of the two sections (rTMS and sham)
  Measurement of sympathetic activity

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Lieh Huang, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital Yunlin Branch, Douliu, Yunlin, Taiwan

IPD SHARING:
Plan to Share IPD: No